CLINICAL TRIAL: NCT05004584
Title: Evaluation of Appetite Measure Visual Analogue Scales in Home-setting: VASA-home
Brief Title: Validation of Appetite Method Visual Analogue Scales in Home-setting: VASA-home
Acronym: VASA-home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chalmers University of Technology (Other)
Responsible Party: Principal Investigator, Rikard Landberg, Head of division of Food and Nutrition Science, Professor Rikard Landberg,, Chalmers University of Technology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 28220086
Record Dates: First submitted 2021-07-16; First posted 2021-08-13 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Overweight and Obesity; Appetitive Behavior
Keywords: Visual analogue scale (VAS); Continuous glucose monitors (CGM)
MeSH Terms: conditions — Overweight; Obesity; Appetitive Behavior | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Wheat home-based (Experimental)
  Interventions: Other: Wheat home-based appetite assessment
- Rye home-based (Experimental)
  Interventions: Other: Rye home-based appetite assessment
- Rye clinic-based (Experimental)
  Interventions: Other: Rye clinic-based appetite assessment
- Wheat clinic-based (Experimental)
  Interventions: Other: Wheat clinic-based appetite assessment
- Wheat/Rye clinic-based with blood sampling (Experimental)
  Interventions: Other: Rye/Wheat clinic-based appetite assessment with blood sampling

INTERVENTIONS:
Other: Wheat home-based appetite assessment — Home-based appetite assessment with diet based on wheat cereal products.
  Arms: Wheat home-based
Other: Rye home-based appetite assessment — Home-based appetite assessment with diet based on rye cereal products.
  Arms: Rye home-based
Other: Wheat clinic-based appetite assessment — Clinic-based appetite assessment with diet based on wheat cereal products.
  Arms: Wheat clinic-based
Other: Rye clinic-based appetite assessment — Clinic-based appetite assessment with diet based on rye cereal products.
  Arms: Rye clinic-based
Other: Rye/Wheat clinic-based appetite assessment with blood sampling — Clinic-based appetite assessment with diet based on rye or wheat cereal products and continuous blood sampling.
  Arms: Wheat/Rye clinic-based with blood sampling

SUMMARY:
The overall aim is to investigate whether there is a difference between methods when a standardized visual analogue scale is used to measure appetite in the home-setting compared to a monitored clinical setting. Furthermore, the intention is to investigate differences in appetite response between diets based on rye or wheat products, as well as the effects on postprandial metabolic response to such diets. Lastly, the effect of venous blood collection on subjective appetite response will be evaluated.

DETAILED DESCRIPTION:
A human dietary intervention study will be conducted at clinical facilities in Gothenburg. The study will be a randomized crossover trial where 30 overweight, but healthy men and women will be recruited. The overall aim is to investigate whether there is a difference between methods when a standardized visual analogue scale (VAS) is used to measure appetite in the home-setting compared to a monitored clinical setting. Furthermore, the intention is to investigate difference in appetite response between diets based on rye or wheat products, as well as the effects on postprandial metabolic response to such diets. Lastly, the effect of venous blood collection on subjective appetite response will be evaluated.

Participants will be complete 3 clinic-based appetite assessments and 2 home-based appetite assessments in random order. The intervention diets will include a fixed amount of rye or wheat cereal products (approx. 650 kcal) as part of a hypocaloric diet with 500 kcal deficit, irrespective of energy requirements of the individual. Participants will follow a standardized meal plan, incorporating intervention products according to their allocation. The meal plan will consist of a breakfast consisting of puffs with milk. The lunch will consist of tomato soup with crisp bread and cheese/jam, and afternoon snack will consist of crisp bread with cheese/jam. Finally, the dinner will consist of goulash soup with soft or crisp bread and jam/cheese. The participants will be provided with all foods needed for this meal plan. During the day participants will need to answer questions about their appetite every 30 minutes from 8:00 to 12:00 and every 60 minutes from 13:00 to 21:00. These questionnaires with VAS will provide data for the comparison of home-setting and monitored clinical setting as well as appetite response between diets.

One out of the three clinic-based assessment days will include continues blood sampling throughout the day allowing evaluation of subjective appetite response on venous blood collection. Also, blood samples will be analyzed for concentration of appetite regulating hormones; glucagon-like peptide-1 (GLP-1), cholecystokinin (CCK) and ghrelin. Furthermore, insulin and triglyceride concentration will be measured as well as exploratory analysis of metabolome, short chain fatty acids (SCFA), epigenetics and gene expression analyses. Baseline fecal samples will be collected and analyzed for composition of the gut microbiome as well as short chain fatty acids (SCFA). Participants will wear a so-called continuous glucose monitors CGM allowing analysis of postprandial blood glucose throughout all 5 appetite assessment days. Measurement of physical activity will be done using Acti-Watches throughout the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age 30-70 years
* Body mass index (BMI) 27-35 kg/m2
* Hemoglobin ≥117g/l for women and for men ≥134g/l
* Thyroid stimulating hormone (TSH) ≤4.30 mIU/L
* Low density lipoprotein (LDL) cholesterol ≤5.30 mmol/L
* Triglycerides ≤2.60 mmol/L
* Signed informed consent
* Having a mobile device, laptop or similar with internet connection. As well as an email, that they are willing to use for answering questions online, both at the clinic and at home.

Exclusion Criteria:

* Blood donation or participation in a clinical study with blood sampling within 30 days prior to screening visit and throughout the study
* Using nicotine products on a daily basis (incl. chewing gum, patches, snus etc.)
* Using e-cigarettes (regardless of nicotine content)
* Following any weight reduction program or having followed one during the last 6 months prior to screening.
* Diastolic blood pressure ≥ 105 mm Hg at screening
* Systolic blood pressure ≥ 160 mm at screening
* History of stomach or gastrointestinal conditions (Inflammatory bowel disease, Crohn's disease, malabsorption, colostomy, bowel resection, gastric bypass surgery etc.)
* More than 10 hours physical activity per week (e.g. sport, fitness or similar).
* History of heart failure or heart attack within 1 year prior to screening
* Having type-I diabetes
* Receiving pharmacological treatment for type-II diabetes
* Previous gastrointestinal surgery, with the exception of minor surgeries such removal of appendix or gall bladder at least 6 months prior to screening.
* Thyroid disorder
* History of drug or alcohol abuse
* Stroke or transient ischemic attack (TIA) within 1 year prior to screening
* Consumption of drugs aimed at weight management or drugs affecting body weight to a degree that is considered unsuitable for study participation by responsible physician.
* Pregnant, lactation or planning a pregnancy within the timeframe of the study. Pregnancy must have ended at least 6 months prior to screening, and lactation must have ended at least 1 month prior to screening.
* Food allergies, intolerances or dietary restrictions (e.g. vegetarian) preventing consumption of any products included in the study
* Unable to sufficiently understand written and spoken Swedish to provide written consent and understand information and instructions from the study personal.
* Lack of suitability for participation in the study, for any reason, as judged by the medical doctor or PI.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2021-11-16 (Actual)

PRIMARY OUTCOMES:
Appetite assessment: hunger | Throughout the appetite assessment days ,13 hours.
  Appetite will be measured through visual analogue scales 1-100mm, filled in by the participants throughout the assessment days.
Appetite assessment: fullness | Throughout the appetite assessment days ,13 hours.
  Appetite will be measured through visual analogue scales 1-100mm, filled in by the participants throughout the assessment days.
Appetite assessment: desire to eat | Throughout the appetite assessment days ,13 hours.
  Appetite will be measured through visual analogue scales 1-100mm, filled in by the participants throughout the assessment days.

SECONDARY OUTCOMES:
Body weight | Through study completion, an average of 5 weeks.
  Body weight is measured after an overnight fast.
Height | Height is measured at baseline.
  The participant is measured to the nearest 0.5 cm without shoes.
Continuous glucose measurement | Throughout the appetite assessment days ,13 hours.
  Interstitial blood glucose will be measured continuously throughout the intervention with so called continuous glucose monitors CGM, and glucose data for all 5 appetite assessment days will be analyzed.
Physical activity | Throughout the appetite assessment days ,13 hours.
  Physical activity will be measured throughout the intervention using Acti-Watches.
Postprandial glucose response | Throughout the appetite assessment days ,13 hours.
  Postprandial blood samples will be analyzed.
Gut microbiome | Gut microbiome is measured at baseline.
  Fecal samples will be collected and analyzed for composition of the gut microbiome
Effect of continous blood sampling on subjective appetite response | Throughout the appetite assessment days ,13 hours.
  Appetite assessment measured through visual analogue scales will be compared between testdays at the clinic with and without continuous blood sampling.
Investigate differences in appetite response between rye- and wheat-based diets | Throughout the appetite assessment days ,13 hours.
  Appetite will be measured through visual analogue scales 1-100mm and scores from rye-based diets and wheat-based diets will be compared.
Insulin | Throughout the appetite assessment days ,13 hours.
  Postprandial blood samples will be analyzed.
Glucagon-like peptide-1 (GLP-1) | Throughout the appetite assessment days ,13 hours.
  Postprandial blood samples will be analyzed.
Ghrelin | Throughout the appetite assessment days ,13 hours.
  Postprandial blood samples will be analyzed.
Cholecystokinin (CCK) | Throughout the appetite assessment days ,13 hours.
  Postprandial blood samples will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Rikard Landberg, Dr, Principal Investigator — Chalmers University of Technology
Locations (1):
- University of Gothenburg, Department of Food and Nutrition and Sport Science, Gothenburg, Sweden

REFERENCES:
- [Derived] Aberg S, Webb DL, Nordin E, Hellstrom PM, Landberg R. Postprandial Effects of Four Test Meals Containing Wholegrain Rye or Refined Wheat Foods on Circulating Incretins, Ghrelin, Glucose, and Inflammatory Markers. J Nutr. 2025 Jan;155(1):185-196. doi: 10.1016/j.tjnut.2024.10.046. Epub 2024 Nov 6. PMID 39515756